CLINICAL TRIAL: NCT04510584
Title: Halting Early Advancement of Residual Disease by Treatment With Bevacizumab and Atezolizumab in Ovarian Cancer
Brief Title: Maintenance Treatment With Bevacizumab and Atezolizumab for Ovarian Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: 19 patients screenfailed, stopping recruitment before first patient enrollment to analyze pilot results from screening samples.
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEARTBEAT-OV; 20-5562 (Other: University Health Network)
Record Dates: First submitted 2020-08-09; First posted 2020-08-12 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Endometrioid Tumor; Fallopian Tube Cancer; Primary Peritoneal Cancer; TP53 Mutation
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atezolizumab and Bevacizumab (Experimental): A cycle will be every 3 weeks.
  Atezolizumab will be given intravenously (by vein) at a dose of 1200 mg once every cycle. Bevacizumab will be given intravenously at a dose of 15 mg/kg once every cycle. Up to 17 cycles of study treatment may be given.
  Participants may be able to receive the study treatment for more than 17 cycles if the participants and the study doctor thinks that they are benefiting.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is a humanized immunoglobulin (IgG1) monoclonal antibody that targets programmed death-ligand 1 (PD-L1) on tumor-infiltrating immune cells (ICs) or tumor cells (TCs) and prevents interaction with the programmed death-1 (PD-1) receptor and B7.1 (CD80), both of which function as inhibitory receptors expressed on T cells and other immune cells.
  Other Names: TECENTRIQ
Drug: Bevacizumab — Bevacizumab is a recombinant humanized IgG1 monoclonal antibody that binds VEGF, a secreted factor that stimulates angiogenesis. Bevacizumab prevents the interaction of VEGF with its receptors and neutralizes the biological activity of VEGF.
  Other Names: AVASTIN

SUMMARY:
This study is being done to look at the combination of the drugs atezolizumab and bevacizumab as a maintenance treatment (treatment given after the main treatment to keep the cancer from coming back or worsening) following standard therapy in patients with high grade ovarian, fallopian tube, or primary peritoneal cancer with a mutation (change) in a gene called TP53. Genes are molecules in the body that are made up of deoxyribonucleic acid (DNA) and control how the body's cells behave.

DETAILED DESCRIPTION:
Atezolizumab and bevacizumab are a type of drug called a monoclonal antibody. Antibodies are proteins that are naturally found in the blood stream that fight infections. A monoclonal antibody is a special kind of antibody that is created in a laboratory that seeks out specific proteins in the body that may be involved in cancers to stop tumor growth.

When tumor cells start to die, broken down pieces of the tumor's DNA gets released into the blood stream, called circulating tumor DNA (ctDNA). Looking at ctDNA may be useful in determining whether the cancer is responding to treatment.

The purpose of this research study is to see whether looking at tumor DNA circulating in the bloodstream can help to determine which patients may respond to atezolizumab and bevacizumab and whether this drug combination is useful, when given as a maintenance treatment for patients with TP53 mutant ovarian, fallopian tube, or primary peritoneal cancer.

ELIGIBILITY:
Inclusion Criteria:

Pre-screening:

* Patients must have histologically confirmed TP53-mutant high grade serous or high grade endometrioid ovarian, fallopian tube, primary peritoneal cancer.
* Ability to understand and the willingness to sign a written Pre-screening Informed consent document.
* Patients must be receiving standard therapy for recurrent disease and have completed 3 cycles of platinum-based chemotherapy, with clinical benefit (in opinion of investigator). Patients with stable disease (in opinion of investigator) after 3 cycles of chemotherapy will also be eligible for pre-screening. There is no limitation on the number of prior lines of therapy. May have received prior PARP-inhibitor therapy or prior bevacizumab or biosimilar.
* Formalin fixed, paraffin embedded (FFPE) tumour sample from the primary cancer must be available.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patients must have a life expectancy ≥16 weeks

Main Study:

* Patients must have histologically confirmed TP53-mutant high grade serous or high grade endometrioid ovarian, fallopian tube, primary peritoneal cancer.
* Must have completed standard therapy for recurrent disease including at least 4 cycles of platinum-based chemotherapy with no clinical and radiographic evidence of disease progression on the post-treatment scan or a rising CA-125 level, following completion of standard therapy. Patients with stable disease and in response (as per Investigators opinion) following completion of chemotherapy will also be eligible for this study. There is no limitation on the number of prior lines of therapy.
* Following completion of platinum-based chemotherapy, patients must have residual disease detectable by TP53 ctDNA
* May have received prior PARP-inhibitor therapy or prior bevacizumab.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Patients must have a life expectancy ≥16 weeks
* Patients must have normal organ and marrow function
* Ongoing prior toxicities related to previous treatments must be recovered to ≤ grade 2 at the time of registration
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must receive first dose of study treatment within 8 weeks after their last dose of platinum based chemotherapy (last dose is the day of the last infusion)
* Postmenopausal or evidence of non-childbearing status for women of childbearing potential. Female patients of childbearing potential should use highly effective contraception and take active measures to avoid pregnancy while undergoing atezolizumab treatment and for at least 5 months after the last dose.
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations
* Formalin fixed, paraffin embedded (FFPE) tumor sample from the primary cancer must be available.
* Pre-treatment CA-125 measurements must meet specific criterion

Exclusion Criteria:

Pre-screening:

* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, or atezolizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, or psychiatric illness/social situations that (in the opinion of Investigator) would limit compliance with study requirements.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1.

Main Study:

* Patients who are receiving any other investigational agents or on-going chemotherapy.
* History of severe allergic reactions attributed to compounds of similar chemical or biologic composition to bevacizumab, or atezolizumab
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active severe infection, symptomatic congestive heart failure, or psychiatric illness/social situations that (in the opinion of Investigator) would limit compliance with study requirements.
* History of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to day 1.
* Invasive procedures defined as follows:

  * Major surgical procedure or significant traumatic injury within 28 days prior to Day 1 therapy, or open biopsy within 28 days prior to Day 1 therapy
  * Anticipation of need for major surgical procedures during the course of the study
* Significant vascular disease within 6 months prior to Day 1
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because of the possible increased risk of bleeding if treatment with antiangiogenic agents is provided.
* Inadequately controlled hypertension, history of cerebrovascular accident, myocardial infarction or unstable angina, serious or inadequately controlled cardiac arrhythmia within 6 months.
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies.
* Resting ECG with QTcF > 470 msec or family history of long QT syndrome.
* History of bowel obstruction within 28 days from proposed start of treatment.
* History or evidence of arterial thrombotic or hemorrhagic disorders within 3 months before proposed start of treatment, non-healing wound, ulcer, or bone fracture.
* Known active HIV or hepatitis B or C infection
* Other malignancy within the last 3 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), Stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for ≥5 years. Patients with a history of localised breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients should be excluded if they have had prior treatment with anti-CTLA-4 antibody or any other antibody or drug specifically targeting T-cell co-stimulation. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 is not allowed.
* The patient has experienced any of the following:

  * The patient has radiographic evidence of cavitating pulmonary lesion(s).
  * The patient has tumour invading or encasing any major blood vessels.
  * The patient has evidence of tumour invading the GI tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumour within 28 days before the first dose of study treatment
  * Patient with extensive pelvic mass at risk of fistulization, or history
  * Active peptic ulcer disease within 28 days before the first dose of study treatment.
  * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
  * Malabsorption syndrome
  * Other disorders associated with a high risk of fistula formation including PEG tube placement.
* Clinically significant gastrointestinal bleeding within 6 months before the first dose of study treatment
* Administration of a live vaccine within 4 weeks prior to start of protocol therapy.
* Patients with diagnosis of immunodeficiency or who are receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The following are exceptions to this exclusion criteria: intranasal, inhaled, topical steroids, or local steroids injections (e.g. intra-articular injection); systemic corticosteroids at physiologic dose not to exceed 10 mg/day of prednisone or equivalent; steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
* History of autoimmune disease, such as, but not restricted to: rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematous, ankylosing spondylitis, scleroderma, or multiple sclerosis requiring treatment within the last two years. Patients with vitiligo or diabetes are not excluded. Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Patients with recent history of thyroiditis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2023-02-22 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Number of participants where increase in circulating deoxyribonucleic acid (ctDNA) level is related to progression | 3 months

SECONDARY OUTCOMES:
Disease free survival rate | 6 months
Disease free survival rate | 12 months
Progression free survival rate | 1 year
Progression free survival rate | 2 years
Number of participants with disease free survival with change from detectable to undetectable TP53 ctDNA | 6 months
Number of participants with disease free survival with change from detectable to undetectable TP53 ctDNA | 12 months
Number of participants with adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Lheureux, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No